CLINICAL TRIAL: NCT02609048
Title: A 12-week, Double-blind, Randomized, Placebo-controlled, Phase 2 Study, to Evaluate the Effects of Two Doses of MBX-8025 in Subjects With Primary Biliary Cirrhosis (PBC) and an Inadequate Response to Ursodeoxycholic Acid (UDCA)
Brief Title: Study to Evaluate the Effects of Two Doses of Seladelpar (MBX-8025) in Subjects With Primary Biliary Cirrhosis (PBC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped early after review of safety and efficacy demonstrated efficacy proof-of-concept and need for dose reduction.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB8025-21528; 2015-002698-39 (EudraCT Number)
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Primary Biliary Cirrhosis (PBC)
Keywords: PBC
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — (2-methyl-4-(5-methyl-2-(4-trifluoromethyl-phenyl)-2H-(1,2,3)triazol-4-ylmethylsulfanyl)phenoxy)acetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo Dose (Placebo Comparator): Participants received 2 placebo-to-match (PTM) seladelpar capsules, orally, once daily for 12 weeks.
  Interventions: Drug: Placebo Comparator
- Seladelpar 50 mg Dose (Experimental): Participants received seladelpar 50 mg capsule (1 x 50 mg capsule) and a PTM seladelpar capsule, orally, once daily for 12 weeks.
  Interventions: Drug: Placebo Comparator; Drug: Experimental: Seladelpar 50 mg
- Seladelpar 200 mg Dose (Experimental): Participants received seladelpar 200 mg capsules (2 x 100 mg capsules), orally, once daily for 12 weeks.
  Interventions: Drug: Experimental: Seladelpar / MBX-8025 200 mg

INTERVENTIONS:
Drug: Placebo Comparator — Placebo Capsule
  Other Names: Placebo
  Arms: Placebo Dose; Seladelpar 50 mg Dose
Drug: Experimental: Seladelpar 50 mg — Seladelpar 50 mg capsule
  Other Names: MBX-8025; Livdelzi®
  Arms: Seladelpar 50 mg Dose
Drug: Experimental: Seladelpar / MBX-8025 200 mg — Seladelpar 100 mg capsules
  Other Names: MBX-8025; Livdelzi®
  Arms: Seladelpar 200 mg Dose

SUMMARY:
The primary objective of this study is to evaluate the effect of seladelpar (MBX-8025) on alkaline phosphatase (AP) levels in participants with primary biliary cirrhosis (PBC).

DETAILED DESCRIPTION:
Primary:

To evaluate the effect of MBX-8025 on Alkaline Phosphatase (AP) levels

Secondary:

To evaluate the safety and tolerability of MBX-8025 in subjects with Primary Biliary Cirrhosis (PBC) To evaluate the effects of MBX-8025 on Primary Biliary Cirrhosis (PBC) response criteria To evaluate the effects of MBX-8025 on other markers of liver function, lipids, pruritus and Quality of Life (QoL)

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated) and any authorizations required by local law
2. 18 to 75 years old (inclusive)
3. Male or female with a diagnosis of PBC, by at least two of the following criteria:

   * History of AP above upper limit of normal (ULN) for at least six months
   * Positive Anti-Mitochondrial Antibodies (AMA) titers (>1/40 on immunofluorescence or M2 positive by enzyme linked immunosorbent assay (ELISA) or positive PBC-specific antinuclear antibodies
   * Documented liver biopsy result consistent with PBC
4. On a stable and recommended dose of UDCA for the past twelve months
5. AP ≥ 1.67 × ULN
6. For females of reproductive potential, use of at least one barrier contraceptive and a second effective birth control method during the study and for at least two weeks after the last dose. For male subjects, use of appropriate contraception (e.g., condoms), so their female partners of reproductive potential do not become pregnant during the study and for at least two weeks after the last dose

Exclusion Criteria:

1. A medical condition, other than PBC, that in the investigator's opinion would preclude full participation in the study or confound its results (e.g., cancer on active treatment)
2. Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) > 3 × ULN
3. Total bilirubin > 2 × ULN
4. Auto-immune hepatitis
5. Primary sclerosing cholangitis
6. Known history of alpha-1-Antitrypsin deficiency
7. Known history of chronic viral hepatitis
8. Creatine kinase above ULN
9. Serum creatinine above ULN
10. For females, pregnancy or breast-feeding
11. Use of colchicine, methotrexate, azathioprine, or systemic steroids in the two months preceding screening
12. Current use of fibrates, including fenofibrates, or simvastatin
13. Use of an experimental treatment for PBC
14. Use of experimental or unapproved immunosuppressant
15. Any other condition(s) that would compromise the safety of the subject or compromise the quality of the clinical study, as judged by the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pol F Boudes, M.D., Study Chair — Gilead Sciences
Locations (49):
- United States (21):
  - Mayo Clinic of Arizona, Phoenix, Arizona
  - University of California, Davis Medical Center, Sacramento, California
  - University of Florida, Gainesville, Florida
  - University of Miami, Center for Liver Diseases, Miami, Florida
  - Norman Gitlin, MD, Atlanta, Georgia
  - Digestive Helathcare of Georgia, Atlanta, Georgia
  - Indiana University Hospital - Clinical Research Center, Indianapolis, Indiana
  - Henry Ford Health System, Detroit, Michigan
  - Gastroenterology Associates of Western Michigan, PLC, d.b.a. West Michigan Clinical Research, Wyoming, Michigan
  - Kansas City Gastroenterology and Hepatology, Kansas City, Missouri
  - St. Louis University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center / The Nebraska Medical Center, Omaha, Nebraska
  - North Shore-Long Island Jewish Health System / Division of Gastroenterology, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai - The Mount Sinai Medical Center, New York, New York
  - Consultants for Clinical Research, Cincinnati, Ohio
  - CHI St. Luke's Health Baylor College of Medicine Medical Center - Advanced Liver Therapies, Houston, Texas
  - Pinnacle Clinical Research, Live Oak, Texas
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas
  - Bon Secours St. Mary's Hospital of Richmond, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
- Canada (2):
  - University of Calgary Liver Unit (Heritage Medical Research Clinic), Calgary, Alberta
  - Toronto General Hospital, Toronto, Ontario
- Germany (15):
  - Charite Universitatsmedizin Berlin - Campus Mitte, Berlin
  - Leber- und Studienzentrum am Checkpoint, Berlin
  - Universitatsklinikum Bonn, Bonn
  - Universitatsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - University Hospital Erlangen, Erlangen
  - Universitatsklinikum Essen, Zentrum fur Innere Medizin, Essen
  - Ifi-Studien und Projekte GmbH, A.d. Asklepios Klinik St. Georg, Hamburg
  - Universitatsklinikum Hamburg-Eppendorf MARTINISTRASSE 52, Hamburg
  - Med. Hochschule Hannover, Klinik fur Gastroenterologie, Hanover
  - Medizinische Universitatsklinik, Heidelberg
  - Gastroenterologische Gemeinschaftspraxis Herne, Herne
  - UKSH, Campus Kiel, Klinik fur Allgemeine Innere Medizin 1, Kiel
  - UKSH, Campus Kiel, Kiel
  - Universitatsklinikum Leipzig AOR, Leipzig
  - Universitatsmedizin der Johannes Gutenberg - Universitat Mainz, Mainz
- Poland (5):
  - Wojewodzki Szpital Obserwacyjno-Zakazny im. Tadeusza w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - SPZOZ Szpital Uniwersytecki w Krakowie, Krakow, Malopolski
  - Centrum Onkologii-Instytut Im. Marii Sklodowskiej-Curie, Warsaw, Masovian Voivodeship
  - SP CSK im. Prof. K. Gibinskiego SUM w Katowicach, Katowice, Silesian Voivodeship
  - ID Clinic Arkadiusz Pisula, Mysłowice, Silesian Voivodeship
- United Kingdom (6):
  - Derriford Hospital, Plymouth, England
  - University Hospital Birmingham NHS Foundation Trust, Birmingham
  - Addenbrooke Hospital, Cambridge
  - Hull and East Yorkshire NHS Trust, Hull
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham

REFERENCES:
- [Derived] Jones D, Boudes PF, Swain MG, Bowlus CL, Galambos MR, Bacon BR, Doerffel Y, Gitlin N, Gordon SC, Odin JA, Sheridan D, Worns MA, Clark V, Corless L, Hartmann H, Jonas ME, Kremer AE, Mells GF, Buggisch P, Freilich BL, Levy C, Vierling JM, Bernstein DE, Hartleb M, Janczewska E, Rochling F, Shah H, Shiffman ML, Smith JH, Choi YJ, Steinberg A, Varga M, Chera H, Martin R, McWherter CA, Hirschfield GM. Seladelpar (MBX-8025), a selective PPAR-delta agonist, in patients with primary biliary cholangitis with an inadequate response to ursodeoxycholic acid: a double-blind, randomised, placebo-controlled, phase 2, proof-of-concept study. Lancet Gastroenterol Hepatol. 2017 Oct;2(10):716-726. doi: 10.1016/S2468-1253(17)30246-7. Epub 2017 Aug 14. PMID 28818518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Canada, Germany, the United Kingdom, and the United States.
Pre-assignment Details: 70 participants were screened.
Groups:
- Seladelpar 200 mg: Participants received seladelpar 200 mg capsules (2 x 100 mg capsules), orally, once daily for 12 weeks.
- Seladelpar 50 mg: Participants received seladelpar 50 mg capsule (1 x 50 mg capsule) and a placebo-to-match (PTM) seladelpar capsule, orally, once daily for 12 weeks.
- Placebo: Participants received 2 PTM seladelpar capsules, orally, once daily for 12 weeks.
Period: Overall Study
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Started | 13 | 14 | 14
Completed | 2 | 4 | 4
Not Completed | 11 | 10 | 10
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Randomized but never treated | 1 | 1 | 1
Not completed — Withdrawal of informed consent | 1 | 0 | 0
Not completed — Reason not specified | 6 | 9 | 9

BASELINE CHARACTERISTICS:
Population: The Safety Population was defined as any randomized participant who received at least 1 dose of medication.
Groups:
- Seladelpar 50 mg: Participants received seladelpar 50 mg capsule (1 x 50 mg capsule) and a PTM seladelpar capsule, orally, once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo | Total
Number analyzed (Participants) | 12 | 13 | 13 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 12 | 33
  >=65 years | 3 | 1 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11.4) | 54 (7.4) | 55 (10.1) | 55 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 12 | 36
  Male | 0 | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 12 | 13 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: For Race, data was not collected for 1 participant in the Seladelpar 50 mg group.
  Participants
    number analyzed (Participants) | 12 | 12 | 13 | 37
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 2 | 0 | 0 | 2
    White | 10 | 12 | 13 | 35
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 5 | 6 | 17
  United Kingdom | 2 | 4 | 3 | 9
  Germany | 3 | 2 | 3 | 8
  Canada | 1 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Baseline Alkaline Phosphatase (AP) Levels
Description: Baseline for AP level was defined as the mean between assessments at Visit 1 (Week -4 to Week 0) and Visit 2 (Week 0).
Time Frame: Baseline
Population: The modified intent-to-treat (mITT) Analysis Set was defined as any randomized participant who received at least 1 dose of medication and had at least 1 on-treatment AP evaluation.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Groups:
- Placebo: Participants received 2 placebo to match (PTM) seladelpar capsules, orally, once daily for 12 weeks.
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 12
units per liter (U/L) | 248.3 (88.69) | 311.6 (94.83) | 232.8 (72.51)

2. Primary Outcome: Percent Change From Baseline in Alkaline Phosphatase (AP) Levels
Description: Percent change in AP serum levels from Baseline to the end of treatment was analyzed. For missing postbaseline data, the last non-missing postbaseline value on treatment was carried forward, with missing assessments imputed by last observation carried forward (LOCF). Baseline for AP level was defined as the mean between assessments at Visit 1 (Week -4 to Week 0) and Visit 2 (Week 0).
Time Frame: Baseline, Week 12
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in AP levels
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 12
percent change in AP levels | -62.83 (4.312) | -53.21 (3.961) | -1.84 (4.020)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — Difference in mean,p-value, and CIs estimated by comparing Seladelpar level with placebo by ANCOVA model.Treatment group as factor,baseline AP assessment as covariate,and percent change from baseline as response variable; Difference in LSM = -60.99, 95% CI 2-sided [-72.85 to -49.13], Standard Error of Mean 5.814
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — Difference in mean,p-value, and confidence intervals (CIs) estimated by comparing Seladelpar level with placebo by ANCOVA model.Treatment group as factor,baseline AP assessment as covariate,and percent change from baseline as response variable; Difference in Least Squares Mean (LSM) = -51.37, 95% CI 2-sided [-63.30 to -39.44], Standard Error of Mean 5.849
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.1167, ANCOVA — Difference in mean,p-value, and CIs estimated by comparing Seladelpar 200 mg versus 50 mg by ANCOVA model.Treatment group as factor,baseline AP assessment as covariate,and percent change from baseline as response variable; Difference in Least Squares Mean (LSM) = -9.62, 95% CI 2-sided [-21.79 to 2.54], Standard Error of Mean 5.963

3. Secondary Outcome: Percentage of Participants With Response as Determined by Composite Endpoint of Alkaline Phosphatase and Total Bilirubin
Description: Participants were defined as responders for the composite endpoint of AP and total bilirubin if their AP level was <1.67 × upper limit of normal (ULN) and had decreased at least 15% from their Baseline level and their total bilirubin value was within the normal range [0.1-1.1 milligrams/deciliter (mg/dL)].
Time Frame: Week 12
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 12
percentage of participants | 100 | 69.2 | 8.3
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p < 0.0001, Fisher Exact — The p-values were calculated from Fisher's exact test comparing each Seladelpar group with Placebo separately
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.0036, Fisher Exact — The p-values were calculated from Fisher's exact test comparing each Seladelpar group with Placebo separately
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.1045, Fisher Exact — The p-values were calculated from Fisher's exact test comparing Seladelpar 200mg versus 50 mg

4. Secondary Outcome: Percent Change From Baseline in Aspartate Aminotransferase (AST)
Description: Percentage change in AST levels from Baseline to the end of treatment was analyzed. For missing postbaseline data, the last non-missing postbaseline value on treatment was carried forward, with missing assessments imputed by LOCF. Baseline for AST level was defined as the last non-missing assessments prior to or on the date of the first study dose.
Time Frame: Baseline, Week 12
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in AST levels
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 12
percent change in AST levels | 232.69 (77.409) | 130.81 (66.933) | -2.02 (69.364)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.0322, ANCOVA — Difference between means, p-value, and CIs are estimated by comparing each Seladelpar level with placebo using ANCOVA model.Treatment group as factor, baseline AST assessment as covariate,and percent change from baseline in AST as response variable; Difference in LSM = 234.71, 95% CI 2-sided [21.28 to 448.14], Standard Error of Mean 104.647
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.1764, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Difference in LSM = 132.82, 95% CI 2-sided [-63.00 to 328.65], Standard Error of Mean 96.015
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.3326, ANCOVA — Difference between means, p-value, and CIs are estimated by comparing Seladelpar 200 mg versus 50 mg using ANCOVA model.Treatment group as factor, baseline AST assessment as covariate, and percent change from baseline in AST as response variable; Difference in LSM = 101.88, 95% CI 2-sided [-109.21 to 312.98], Standard Error of Mean 103.504

5. Secondary Outcome: Percent Change From Baseline in Alanine Aminotransferase (ALT)
Description: Percentage change in ALT levels from Baseline to the end of treatment was analyzed. For missing postbaseline data, the last non-missing postbaseline value on treatment was carried forward, with missing assessments imputed by LOCF. Baseline for ALT level was defined as the last non-missing assessments prior to or on the date of the first study dose.
Time Frame: Baseline, Week 12
Population: Participants in the mITT analysis set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in ALT levels
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 12
percent change in ALT levels | 181.11 (77.864) | 111.83 (68.061) | -4.67 (69.632)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.0849, ANCOVA — Difference between means,p-value, and CIs are estimated by comparing each Seladelpar level with placebo using ANCOVA model.Treatment group as a factor, baseline ALT assessment as covariate,and percent change from baseline in ALT as response variable; Difference in LSM = 185.78, 95% CI 2-sided [-27.10 to 398.66], Standard Error of Mean 104.379
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.2409, ANCOVA — Difference between means,p-value,and CIs are estimated by comparing each Seladelpar level with placebo using ANCOVA model.Treatment group as a factor,baseline ALT assessment as covariate, and percent change from baseline in ALT as response variable; Difference in LSM = 116.50, 95% CI 2-sided [-82.22 to 315.23], Standard Error of Mean 97.437
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.5154, ANCOVA — Difference between means,p-value,and CIs are estimated by comparing Seladelpar 200 mg versus 50 mg using ANCOVA model.Treatment group as a factor,baseline ALT assessment as covariate, and percent change from baseline in ALT as response variable; Difference in LSM = 69.28, 95% CI 2-sided [-145.47 to 284.03], Standard Error of Mean 105.295

6. Secondary Outcome: Percent Change From Baseline in Gamma-glutamyl Transferase (GGT)
Description: Percentage change in GGT levels from Baseline to the end of treatment was analyzed. For missing postbaseline data, the last non-missing postbaseline value on treatment was carried forward, with missing assessments imputed by LOCF. Baseline for GGT level was defined as the last non-missing assessments prior to or on the date of the first study dose.
Time Frame: Baseline, Week 12
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in GGT levels
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 12
percent change in GGT levels | -47.17 (9.084) | -42.60 (7.796) | -1.83 (7.889)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.0007, ANCOVA — Difference between means, p-value,and CIs are estimated by comparing each Seladelpar level with placebo using ANCOVA model.Treatment group as a factor, baseline GGT assessment as covariate,and percent change from baseline in GGT as response variable; Difference in LSM = -45.34, 95% CI 2-sided [-70.04 to -20.64], Standard Error of Mean 12.112
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.0008, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Difference in LSM = -40.78, 95% CI 2-sided [-63.28 to -18.28], Standard Error of Mean 11.033
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.7155, ANCOVA — Difference between means, p-value,and CIs are estimated by comparing Seladelpar 200 mg versus 50 mg using ANCOVA model.Treatment group as a factor, baseline GGT assessment as covariate,and percent change from baseline in GGT as response variable; Difference in LSM = -4.56, 95% CI 2-sided [-29.85 to 20.73], Standard Error of Mean 12.401

7. Secondary Outcome: Percent Change From Baseline in 5'Nucleotidase (5NT)
Description: Percentage change in 5'Nucleotidase levels from Baseline to the end of treatment was analyzed. For missing postbaseline data, the last non-missing postbaseline value on treatment was carried forward, with missing assessments imputed by LOCF. Baseline for 5NT level was defined as the last non-missing assessments prior to or on the date of the first study dose.
Time Frame: Baseline, Week 12
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in 5'Nucleotidase levels
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 12
percent change in 5'Nucleotidase levels | -34.35 (8.446) | -24.92 (7.148) | -0.08 (7.305)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.0050, ANCOVA — Difference between means,p-value, and CIs are estimated by comparing each Seladelpar level with placebo using ANCOVA model.Treatment group as a factor, baseline 5NT assessment as covariate,and percent change from baseline in 5NT as response variable; Difference in LSM = -34.27, 95% CI 2-sided [-57.40 to -11.14], Standard Error of Mean 11.342
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.0199, ANCOVA — [p-value comment as in outcome 7, analysis 1]; Difference in LSM = -24.84, 95% CI 2-sided [-45.47 to -4.21], Standard Error of Mean 10.116
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.4161, ANCOVA — Difference between means,p-value, and CIs are estimated by comparing Seladelpar 200 mg versus 50 mg using ANCOVA model.Treatment group as a factor, baseline 5NT assessment as covariate,and percent change from baseline in 5NT as response variable; Difference in LSM = -9.43, 95% CI 2-sided [-32.77 to 13.90], Standard Error of Mean 11.442

8. Secondary Outcome: Percent Change From Baseline in Total Bilirubin
Description: Percentage change in total bilirubin levels from Baseline to the end of treatment was analyzed. For missing postbaseline data, the last non-missing postbaseline value on treatment was carried forward, with missing assessments imputed by LOCF. Baseline for total bilirubin level was defined as the last non-missing assessments prior to or on the date of the first study dose.
Time Frame: Baseline, Week 12
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in total bilirubin levels
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 12
percent change in total bilirubin levels | 1.40 (6.384) | -16.79 (5.586) | -4.79 (5.793)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.4780, ANCOVA — Difference between means,p-value, and CIs estimated by comparing each Seladelpar level with placebo by ANCOVA model.Treatment group as factor, baseline assessment as covariate, and percent change from baseline in total bilirubin as response variable; Difference in LSM = 6.20, 95% CI 2-sided [-11.40 to 23.79], Standard Error of Mean 8.626
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.1459, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Difference in LSM = -12.00, 95% CI 2-sided [-28.40 to 4.41], Standard Error of Mean 8.043
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.0407, ANCOVA — Difference between means,p-value, and CIs estimated by comparing Seladelpar 200 mg versus 50 mg by ANCOVA model.Treatment group as factor, baseline assessment as covariate, and percent change from baseline in total bilirubin as response variable; Difference in LSM = 18.19, 95% CI 2-sided [0.82 to 35.57], Standard Error of Mean 8.521

9. Secondary Outcome: Percent Change From Baseline in Conjugated Bilirubin
Description: Percentage change in conjugated bilirubin levels from Baseline to the end of treatment was analyzed. For missing postbaseline data, the last non-missing postbaseline value on treatment was carried forward, with missing assessments imputed by LOCF. Baseline for conjugated bilirubin level was defined as the last non-missing assessments prior to or on the date of the first study dose.
Time Frame: Baseline, Week 12
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in conjugated bilirubin
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 12
percent change in conjugated bilirubin | 42.30 (10.213) | 2.00 (8.932) | 10.84 (9.296)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.0300, ANCOVA — Difference between means,p-value,and CIs are estimated by each Seladelpar level with placebo using ANCOVA model.Treatment group as factor,baseline assessment as covariate,and percent change from baseline in conjugated bilirubin as response variable; Difference in LSM = 31.47, 95% CI 2-sided [3.26 to 59.67], Standard Error of Mean 13.831
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.4979, ANCOVA — [p-value comment as in outcome 9, analysis 1]; Difference in LSM = -8.84, 95% CI 2-sided [-35.11 to 17.44], Standard Error of Mean 12.883
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.0058, ANCOVA — Difference between means,p-value,and CIs are estimated for Seladelpar 200 mg versus 50 mg using ANCOVA model.Treatment group as factor,baseline assessment as covariate,and percent change from baseline in conjugated bilirubin as response variable; Difference in LSM = 40.30, 95% CI 2-sided [12.58 to 68.02], Standard Error of Mean 13.591

10. Secondary Outcome: Percent Change From Baseline in Unconjugated Bilirubin
Description: Percentage change in unconjugated bilirubin levels from Baseline to the end of treatment was analyzed. For missing postbaseline data, the last non-missing postbaseline value on treatment was carried forward, with missing assessments imputed by LOCF. Baseline for unconjugated bilirubin level was defined as the last non-missing assessments prior to or on the date of the first study dose.
Time Frame: Baseline, Week 12
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in unconjugated bilirubin
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 12
percent change in unconjugated bilirubin | -11.86 (6.197) | -23.04 (5.431) | -8.89 (5.620)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.7244, ANCOVA — Difference between means,p-value, and CIs are estimated by comparing Seladelpar level with placebo using ANCOVA model.Treatment group as a factor,baseline assessment as covariate, and percent change from baseline as the response variable; Difference in LSM = -2.97, 95% CI 2-sided [-20.03 to 14.08], Standard Error of Mean 8.362
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.0800, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Difference in LSM = -14.15, 95% CI 2-sided [-30.10 to 1.80], Standard Error of Mean 7.819
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.1874, ANCOVA — Difference between means,p-value, and CIs are estimated by comparing Seladelpar 200 mg versus 50 mg using ANCOVA model.Treatment group as a factor,baseline assessment as covariate, and percent change from baseline as the response variable; Difference in LSM = 11.18, 95% CI 2-sided [-5.73 to 28.08], Standard Error of Mean 8.290

11. Secondary Outcome: Percent Change From Baseline in Bone-specific AP Levels
Description: Percentage change in bone-specific AP levels from Baseline to the end of treatment was analyzed. For missing postbaseline data, the last non-missing postbaseline value on treatment was carried forward, with missing assessments imputed by LOCF. Baseline for bone-specific level was defined as the last non-missing assessments prior to or on the date of the first study dose.
Time Frame: Baseline, Week 12
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in bone-specific AP level
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 12
percent change in bone-specific AP level | -50.39 (4.837) | -39.09 (4.355) | -4.43 (4.544)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — Difference between means,p-value,and CIs are estimated comparing each Seladelpar level with placebo using ANCOVA model.Treatment group as factor,baseline bone-specific AP assessment as covariate,and percent change from baseline as response variable; Difference in LSM = -45.96, 95% CI 2-sided [-59.50 to -32.42], Standard Error of Mean 6.638
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Difference in LSM = -34.66, 95% CI 2-sided [-47.83 to -21.48], Standard Error of Mean 6.460
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.0924, ANCOVA — Difference between means,p-value,and CIs are estimated comparing Seladelpar 200 mg versus 50 mg using ANCOVA model.Treatment group as factor,baseline bone-specific AP assessment as covariate,and percent change from baseline as response variable; Difference in LSM = -11.30, 95% CI 2-sided [-24.58 to 1.97], Standard Error of Mean 6.508

12. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG)
Description: Percentage change in TG levels from Baseline to the end of treatment was analyzed. For missing postbaseline data, the last non-missing postbaseline value on treatment was carried forward, with missing assessments imputed by LOCF. Baseline for TG level was defined as the last non-missing assessments prior to or on the date of the first study dose.
Time Frame: Baseline, Week 12
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in TG levels
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 12
percent change in TG levels | -7.11 (9.415) | -30.27 (8.243) | 7.04 (8.617)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.2777, ANCOVA — Difference between means,p-value, and CIs are estimated by comparing each Seladelpar level with placebo using ANCOVA model.Treatment group as factor, baseline TG assessment as a covariate, and percent change from baseline in TG as response variable; Difference in LSM = -14.15, 95% CI 2-sided [-40.27 to 11.97], Standard Error of Mean 12.807
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.0039, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Difference in LSM = -37.31, 95% CI 2-sided [-61.67 to -12.95], Standard Error of Mean 11.946
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.0734, ANCOVA — Difference between means,p-value, and CIs are estimated by comparing Seladelpar 200 mg versus 50 mg using ANCOVA model.Treatment group as factor, baseline TG assessment as a covariate, and percent change from baseline in TG as response variable; Difference in LSM = 23.16, 95% CI 2-sided [-2.33 to 48.65], Standard Error of Mean 12.498

13. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC)
Description: Percentage change in TC levels from Baseline to the end of treatment was analyzed. For missing postbaseline data, the last non-missing postbaseline value on treatment was carried forward, with missing assessments imputed by LOCF. Baseline for TC level was defined as the last non-missing assessments prior to or on the date of the first study dose.
Time Frame: Baseline, Week 12
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in TC levels
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 12
percent change in TC levels | -16.43 (3.250) | -8.44 (2.774) | -0.32 (2.905)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.0010, ANCOVA — Difference between means,p-value,and CIs are estimated by comparing each Seladelpar level with placebo using ANCOVA model.Treatment group as factor, baseline TC assessment as covariate,and percent change from baseline in TC as the response variable; Difference in LSM = -16.12, 95% CI 2-sided [-25.16 to -7.07], Standard Error of Mean 4.433
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.0504, ANCOVA — [p-value comment as in outcome 13, analysis 1]; Difference in LSM = -8.13, 95% CI 2-sided [-16.27 to 0.02], Standard Error of Mean 3.992
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.0738, ANCOVA — Difference between means,p-value,and CIs are estimated by comparing Seladelpar 200 mg versus 50 mg using ANCOVA model.Treatment group as factor, baseline TC assessment as covariate,and percent change from baseline in TC as the response variable; Difference in LSM = -7.99, 95% CI 2-sided [-16.80 to 0.81], Standard Error of Mean 4.317

14. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C)
Description: Percentage change in HDL-C levels from Baseline to the end of treatment was analyzed. For missing postbaseline data, the last non-missing postbaseline value on treatment was carried forward, with missing assessments imputed by LOCF. Baseline for HDL-C level was defined as the last non-missing assessments prior to or on the date of the first study dose.
Time Frame: Baseline, Week 12
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in HDL-C levels
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 12
percent change in HDL-C levels | -13.06 (4.326) | 3.44 (3.747) | 4.33 (3.884)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.0057, ANCOVA — Difference between means,p-value,and CIs estimated by comparing each Seladelpar level with placebo using ANCOVA model.Treatment group as factor,baseline HDL-C assessment as covariate,and percent change from baseline in HDL-C as response variable; Difference in LSM = -17.39, 95% CI 2-sided [-29.32 to -5.46], Standard Error of Mean 5.848
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.8703, ANCOVA — [p-value comment as in outcome 14, analysis 1]; Difference in LSM = -0.89, 95% CI 2-sided [-11.85 to 10.08], Standard Error of Mean 5.378
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.0076, ANCOVA — Difference between means,p-value,and CIs estimated by comparing Seladelpar 200 mg versus 50 mg using ANCOVA model.Treatment group as factor,baseline HDL-C assessment as covariate,and percent change from baseline in HDL-C as response variable; Difference in LSM = -16.51, 95% CI 2-sided [-28.30 to -4.71], Standard Error of Mean 5.781

15. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C)
Description: Percentage change in LDL-C levels from Baseline to the end of treatment was analyzed. For missing postbaseline data, the last non-missing postbaseline value on treatment was carried forward, with missing assessments imputed by LOCF. Baseline for LDL-C level was defined as the last non-missing assessments prior to or on the date of the first study dose.
Time Frame: Baseline, Week 12
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in LDL-C levels
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 12
percent change in LDL-C levels | -17.63 (4.372) | -12.83 (3.763) | -2.78 (3.958)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.0186, ANCOVA — Difference between means,p-value, and CIs estimated by comparing each Seladelpar level with placebo using ANCOVA model.Treatment group as factor,baseline LDL-C assessment as covariate,and percent change from baseline in LDL-C as response variable; Difference in LSM = -14.85, 95% CI 2-sided [-27.05 to -2.66], Standard Error of Mean 5.981
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.0745, ANCOVA — [p-value comment as in outcome 15, analysis 1]; Difference in LSM = -10.06, 95% CI 2-sided [-21.17 to 1.06], Standard Error of Mean 5.448
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.4131, ANCOVA — Difference between means,p-value, and CIs estimated by comparing Seladelpar 200 mg versus 50 mg using ANCOVA model.Treatment group as factor,baseline LDL-C assessment as covariate,and percent change from baseline in LDL-C as response variable; Difference in LSM = -4.80, 95% CI 2-sided [-16.60 to 7.00], Standard Error of Mean 5.785

16. Secondary Outcome: Number of Participants Who Were Non-responders as Determined by Published PBC Response Criteria (Paris I)
Description: Published criteria for response to treatment in PBC included Paris I criteria. For Paris I, the criteria used to measure the PBC participants' response to study treatment was: AP ≤ 3x ULN and AST ≤ 2x ULN and Total Bilirubin ≤ 1 mg/dL. Participants who satisfied the criteria were defined as responders and those who did not were considered nonresponders if all the elements had non-missing assessments at that visit. The number of nonresponders were reported, the missing assessments were imputed by LOCF.
Time Frame: Week 12
Population: Participants in the mITT Analysis Set with available data were analyzed. Only participants who did not meet the criteria for response at Baseline were included in the analysis. Baseline for published PBC response criteria (Paris I) was defined as the last non-missing assessments prior to or on the date of the first study dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 2 | 4 | 2
Participants | 2 | 2 | 2
Statistical Analysis 1: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.4667, Fisher Exact — Fisher's exact test between each Seladelpar level compared with placebo was used to obtain the p-value
Statistical Analysis 2: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.4667, Fisher Exact — Fisher's exact test between Seladelpar 200 mg versus 50 mg was used to obtain the p-value

17. Secondary Outcome: Number of Participants Who Were Non-responders as Determined by Published PBC Response Criteria (Paris II)
Description: Published criteria for response to treatment in PBC included Paris II criteria. For Paris II, the criteria used to measure the PBC participants' response to study treatment was: AP ≤ 1.5x ULN and AST ≤ 1.5x ULN and Total Bilirubin ≤ 1 mg/dL. Participants who satisfied the criteria were defined as responders and those who did not were considered nonresponders if all the elements had non-missing assessments at that visit. The number of nonresponders were reported, the missing assessments were imputed by LOCF.
Time Frame: Week 12
Population: Participants in the mITT Analysis Set with available data were analyzed. Only participants who did not meet the criteria for response at Baseline were included in the analysis. Baseline for published PBC response criteria (Paris II) was defined as the last non-missing assessments prior to or on the date of the first study dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 8 | 13 | 9
Participants | 5 | 8 | 9
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.0824, Fisher Exact — Fisher's exact test between each Seladelpar level compared with placebo was used to obtain the p-value
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.0537, Fisher Exact — Fisher's exact test between each Seladelpar level compared with placebo was used to obtain the p-value
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 1.0000, Fisher Exact — Fisher's exact test between Seladelpar 200 mg versus 50 mg was used to obtain the p-value

18. Secondary Outcome: Number of Participants Who Were Non-responders as Determined by Published PBC Response Criteria (Toronto I)
Description: Published criteria for response to treatment in PBC included Toronto I criteria. For Toronto I, the criteria used to measure the PBC participants' response to study treatment was: AP ≤ 1.67x ULN. Participants who satisfied the criteria were defined as responders and those who did not were considered nonresponders if all the elements had non-missing assessments at that visit. The number of nonresponders were reported, the missing assessments were imputed by LOCF.
Time Frame: Week 12
Population: Participants in the mITT Analysis Set with available data were analyzed. Only participants who did not meet the criteria for response at Baseline were included in the analysis. Baseline for published PBC response criteria (Toronto I) was defined as the last non-missing assessments prior to or on the date of the first study dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 4 | 11 | 8
Participants | 0 | 3 | 7
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.0101, Fisher Exact — Fisher's exact test between each Seladelpar level compared with placebo was used to obtain the p-value
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.0198, Fisher Exact — Fisher's exact test between each Seladelpar level compared with placebo was used to obtain the p-value
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.5165, Fisher Exact — Fisher's exact test between Seladelpar 200 mg versus 50 mg was used to obtain the p-value

19. Secondary Outcome: Number of Participants Who Were Non-responders as Determined by Published PBC Response Criteria (Toronto II)
Description: Published criteria for response to treatment in PBC included Toronto II criteria. For Toronto II, the criteria used to measure the PBC participants' response to study treatment was: AP ≤ 1.76x ULN. Participants who satisfied the criteria were defined as responders and those who did not were considered nonresponders if all the elements had non-missing assessments at that visit. The number of nonresponders were reported, the missing assessments were imputed by LOCF.
Time Frame: Week 12
Population: Participants in the mITT Analysis Set with available data were analyzed. Only participants who did not meet the criteria for response at Baseline were included in the analysis. Baseline for published PBC response criteria (Toronto II) was defined as the last non-missing assessments prior to or on the date of the first study dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 4 | 11 | 9
Participants | 0 | 2 | 7
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.0101, Fisher Exact — Fisher's exact test between each Seladelpar level compared with placebo was used to obtain the p-value
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.0055, Fisher Exact — Fisher's exact test between each Seladelpar level compared with placebo was used to obtain the p-value
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 1.0000, Fisher Exact — Fisher's exact test between Seladelpar 200 mg versus 50 mg was used to obtain the p-value

20. Secondary Outcome: United Kingdom-Primary Biliary Cirrhosis/Cholangitis (UK-PBC) Risk Score
Description: The UK-PBC Risk Score was used to estimate the risk that a PBC participant would develop liver failure that would require liver transplantation within 5, 10 or 15 years from diagnosis. The UK-PBC Risk Score calculation was adapted based on the AP assessment, transaminases (refers to the ALT, where available, otherwise the AST assessment) and total bilirubin assessment respectively at end of treatment divided by its upper limits of the corresponding normal ranges; "albumin" and "platelet" refer to the baseline values of these parameters divided by their corresponding lower limits of normal ranges. Missing assessments at end of treatment was imputed by last observation carried forward (LOCF). The UK-PBC risk scores for 5, 10 and 15 years was calculated for each treatment group
Time Frame: Week 12
Population: Participants in the mITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage risk
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 12 | 12
percentage risk
  UK-PBC Risk Score by 5 years | 1.3642 (0.95452) | 1.8530 (2.32301) | 3.1102 (5.1892)
  UK-PBC Risk Score by 10 years | 3.9796 (2.74081) | 5.2712 (6.31842) | 8.3004 (12.51699)
  UK-PBC Risk Score by 15 years | 6.4392 (4.36737) | 8.3379 (9.57184) | 12.4804 (17.05244)

21. Secondary Outcome: Change From Baseline in 5-Dimension (5-D) Itch Scale Score
Description: The 5-D itch scale was used to for the multidimensional quantification of pruritus over time. It assessed five aspects of itching: degree, duration, direction, disability, and distribution.The 5-D itch Scale is a measure of itching that has been validated in patients with chronic pruritus to detect changes over time. A 5-D itch scale score typically ranges from 5 to 25 with a higher score indicating greater itch severity, where 5 represents no pruritus (itching) and 25 represents the most severe pruritus; Each dimension is scored separately, and the scores are added together to get a total 5-D itch score. Higher scores indicate worsening of itching. The total 5-D itch Scale score change from Baseline was calculated. Baseline for 5-D itch scale was defined as the last non-missing assessments prior to or on the date of the first study dose. Missing assessments at end of treatment was imputed by LOCF.
Time Frame: Baseline, Week 12
Population: Participants in the mITT Analysis Set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 10 | 13 | 11
score on a scale | -0.9 (1.31) | 0.5 (1.15) | 0.2 (1.25)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.5379, ANCOVA — Difference between means,p-value, and CIs are estimated by comparing each Seladelpar level with placebo using ANCOVA model.Treatment group as factor, baseline score as covariate, and change from baseline score as the response variable; Difference in LSM = -1.1, 95% CI 2-sided [-4.8 to 2.6], Standard Error of Mean 1.82
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.8949, ANCOVA — [p-value comment as in outcome 21, analysis 1]; Difference in LSM = 0.2, 95% CI 2-sided [-3.3 to 3.7], Standard Error of Mean 1.70
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.4431, ANCOVA — Difference between means,p-value, and CIs are estimated by comparing Seladelpar 200 mg versus 50 mg using ANCOVA model.Treatment group as factor, baseline score as covariate, and change from baseline score as the response variable; Difference in LSM = -1.4, 95% CI 2-sided [-4.9 to 2.2], Standard Error of Mean 1.75

22. Secondary Outcome: Change From Baseline in Pruritus Visual Analog Scale (VAS) Score
Description: VAS was used to measure pruritis in participants with PBC. Participants placed a mark representing their level of itching since the previous measurement on a 100-mm VAS with 0 indicating no itching and 100 mm indicating the worst possible itching. Higher scores indicated worsening of itching The change from Baseline was presented by treatment group. Baseline for VAS score was defined as the last non-missing assessments prior to or on the date of the first study dose. Missing assessments at end of treatment was imputed by LOCF.
Time Frame: Baseline, Week 12
Population: Participants in the mITT Analysis Set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 9 | 12 | 12
score on a scale | 0.9 (7.54) | -0.7 (6.35) | 8.3 (6.42)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Test type: Superiority; p = 0.4674, ANCOVA — Difference between means,p-value, and CIs are estimated by comparing each Seladelpar level with placebo using ANCOVA model. Treatment group as factor, baseline score as a covariate, and change from baseline score as the response variable; Difference in LSM = -7.4, 95% CI 2-sided [-28.0 to 13.2], Standard Error of Mean 10.07
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Test type: Superiority; p = 0.3236, ANCOVA — [p-value comment as in outcome 22, analysis 1]; Difference in LSM = -9.0, 95% CI 2-sided [-27.4 to 9.4], Standard Error of Mean 8.99
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Test type: Superiority; p = 0.8723, ANCOVA — Difference between means,p-value, and CIs are estimated by comparing Seladelpar 200 mg versus 50 mg using ANCOVA model. Treatment group as factor, baseline score as a covariate, and change from baseline score as the response variable; Difference in LSM = 1.6, 95% CI 2-sided [-18.7 to 21.9], Standard Error of Mean 9.92

23. Secondary Outcome: Change From Baseline in PBC-40 Quality of Life Questionnaire
Description: The PBC-40 questionnaire was used to evaluate health-related quality of life measures, specifically fatigue. The PBC-40 questionnaire is a disease-specific tool developed to specifically measure the psychometric profile of PBC patients. It consists of 40 items divided into the six domains relevant to PBC including Cognitive, Social, EmotionalFunction, Fatigue, Itch, and Other Symptoms/General Questions. Items are scored from 1 to 5 and individual items scores are summed to give a total domain score. PBC 40 QoL domain score ranges are:Cognitive (6-30), Emotional Function (3-15),Fatigue (11-55), Itch (3-15),Social (10-50),Symptoms (7-35).Higher scores represent high impact and lower scores low impact of PBC on quality of life.The change and percentage change from Baseline for individual domain score at end of treatment were reported. Baseline for PBC-40 questionnaire was the last non-missing assessments prior to or on the date of the first study dose.Missing assessments imputed by LOCF.
Time Frame: Baseline, Week 12
Population: Participants in the mITT Analysis Set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 7 | 11 | 10
score on a scale
  Cognitive Domain Score | 2.6 (0.96) | 0.9 (0.76) | -0.8 (0.80)
  Social Domain Score | 3.2 (1.32) | 0.3 (1.06) | -0.5 (1.09)
  Emotional Function Domain Score | 0.4 (0.73) | 0.4 (0.58) | 0.0 (0.62)
  Fatigue Domain Score | -0.3 (1.50) | 2.3 (1.20) | -1.9 (1.26)
  Itch Domain Score | -0.6 (0.81) | 0.3 (0.65) | -0.4 (0.67)
  Symptoms Domain Score | 1.1 (0.76) | 0.9 (0.62) | -1.5 (0.64)
Statistical Analysis 1: Comparison: Seladelpar 200 mg vs Placebo; Cognitive Domain Score; Test type: Superiority; p = 0.0115, ANCOVA — Difference between means,p-value,and CIs are estimated comparing each Seladelpar level with placebo using ANCOVA model.Treatment group as factor,baseline PBC 40 QoL domain score as covariate, change from baseline in domain score as response variable; Difference in LSM = 3.4, 95% CI 2-sided [0.8 to 6.0], Standard Error of Mean 1.25
Statistical Analysis 2: Comparison: Seladelpar 50 mg vs Placebo; Cognitive Domain Score; Test type: Superiority; p = 0.1256, ANCOVA — [p-value comment as in outcome 23, analysis 1]; Difference in LSM = 1.8, 95% CI 2-sided [-0.5 to 4.0], Standard Error of Mean 1.10
Statistical Analysis 3: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Cognitive Domain Score; Test type: Superiority; p = 0.1842, ANCOVA — Difference between means,p-value,and CIs are estimated comparing Seladelpar 200 mg versus 50 mg using ANCOVA model.Treatment group as factor,baseline PBC 40 QoL domain score as covariate, change from baseline in domain score as response variable; Difference in LSM = 1.7, 95% CI 2-sided [-0.9 to 4.2], Standard Error of Mean 1.22
Statistical Analysis 4: Comparison: Seladelpar 200 mg vs Placebo; Social Domain Score; Test type: Superiority; p = 0.0420, ANCOVA — [p-value comment as in outcome 23, analysis 1]; Difference in LSM = 3.7, 95% CI 2-sided [0.1 to 7.2], Standard Error of Mean 1.70
Statistical Analysis 5: Comparison: Seladelpar 50 mg vs Placebo; Social Domain Score; Test type: Superiority; p = 0.6384, ANCOVA — [p-value comment as in outcome 23, analysis 1]; Difference in LSM = 0.7, 95% CI 2-sided [-2.4 to 3.9], Standard Error of Mean 1.54
Statistical Analysis 6: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Social Domain Score; Test type: Superiority; p = 0.1035, ANCOVA — [p-value comment as in outcome 23, analysis 3]; Difference in LSM = 2.9, 95% CI 2-sided [-0.6 to 6.5], Standard Error of Mean 1.73
Statistical Analysis 7: Comparison: Seladelpar 200 mg vs Placebo; Emotional Function Domain Score; Test type: Superiority; p = 0.6967, ANCOVA — [p-value comment as in outcome 23, analysis 1]; Difference in LSM = 0.4, 95% CI 2-sided [-1.6 to 2.4], Standard Error of Mean 0.96
Statistical Analysis 8: Comparison: Seladelpar 50 mg vs Placebo; Emotional Function Domain Score; Test type: Superiority; p = 0.6164, ANCOVA — [p-value comment as in outcome 23, analysis 1]; Difference in LSM = 0.4, 95% CI 2-sided [-1.3 to 2.2], Standard Error of Mean 0.85
Statistical Analysis 9: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Emotional Function Domain Score; Test type: Superiority; p = 0.9548, ANCOVA; Difference in LSM = -0.1, 95% CI 2-sided [-2.0 to 1.9], Standard Error of Mean 0.93
Statistical Analysis 10: Comparison: Seladelpar 200 mg vs Placebo; Itch Domain Score; Test type: Superiority; p = 0.8286, ANCOVA — [p-value comment as in outcome 23, analysis 1]; Difference in LSM = -0.2, 95% CI 2-sided [-2.4 to 1.9], Standard Error of Mean 1.04
Statistical Analysis 11: Comparison: Seladelpar 50 mg vs Placebo; Fatigue Domain Score; Test type: Superiority; p = 0.0226, ANCOVA — [p-value comment as in outcome 23, analysis 1]; Difference in LSM = 4.2, 95% CI 2-sided [0.6 to 7.8], Standard Error of Mean 1.74
Statistical Analysis 12: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Fatigue Domain Score; Test type: Superiority; p = 0.1861, ANCOVA — [p-value comment as in outcome 23, analysis 3]; Difference in LSM = -2.6, 95% CI 2-sided [-6.6 to 1.4], Standard Error of Mean 1.92
Statistical Analysis 13: Comparison: Seladelpar 200 mg vs Placebo; Fatigue Domain Score; Test type: Superiority; p = 0.4159, ANCOVA — [p-value comment as in outcome 23, analysis 1]; Difference in LSM = 1.6, 95% CI 2-sided [-2.4 to 5.7], Standard Error of Mean 1.96
Statistical Analysis 14: Comparison: Seladelpar 50 mg vs Placebo; Itch Domain Score; Test type: Superiority; p = 0.4848, ANCOVA — [p-value comment as in outcome 23, analysis 1]; Difference in LSM = 0.7, 95% CI 2-sided [-1.3 to 2.6], Standard Error of Mean 0.93
Statistical Analysis 15: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Itch Domain Score; Test type: Superiority; p = 0.4048, ANCOVA — [p-value comment as in outcome 23, analysis 3]; Difference in LSM = -0.9, 95% CI 2-sided [-3.1 to 1.3], Standard Error of Mean 1.05
Statistical Analysis 16: Comparison: Seladelpar 200 mg vs Placebo; Symptoms Domain Score; Test type: Superiority; p = 0.0141, ANCOVA — [p-value comment as in outcome 23, analysis 1]; Difference in LSM = 2.6, 95% CI 2-sided [0.6 to 4.7], Standard Error of Mean 1.00
Statistical Analysis 17: Comparison: Seladelpar 50 mg vs Placebo; Symptoms Domain Score; Test type: Superiority; p = 0.0138, ANCOVA — [p-value comment as in outcome 23, analysis 1]; Difference in LSM = 2.4, 95% CI 2-sided [0.5 to 4.2], Standard Error of Mean 0.90
Statistical Analysis 18: Comparison: Seladelpar 200 mg vs Seladelpar 50 mg; Symptoms Domain Score; Test type: Superiority; p = 0.7911, ANCOVA — [p-value comment as in outcome 23, analysis 3]; Difference in LSM = 0.3, 95% CI 2-sided [-1.8 to 2.3], Standard Error of Mean 0.98

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to 16.4 weeks; Adverse events: Up to 14.7 weeks
Description: All-cause mortality: All Randomized Analysis Set included participants who were randomized in the study; Adverse events: The Safety Analysis Set included randomized participants who received at least 1 dose of medication.
Arm/Group | Seladelpar 200 mg | Seladelpar 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 10/12 | 11/13 | 10/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Seladelpar 200 mg (N=12) | Seladelpar 50 mg (N=13) | Placebo (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 1 | 0
Transaminases increased (Investigations) | 1 | 1 | 0
Urine output increased (Investigations) | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Lichenification (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Because the study was discontinued before its completion, the interpretation of the results is limited by the small sample size and some imbalance in baseline characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years